CLINICAL TRIAL: NCT02070523
Title: Pegylated Liposomal Doxorubicin-contained Versus Daunorubicin-contained VDCLD Regimen in Previously Untreated Adult Patients With Acute Lymphoblastic Leukemia: Complete Remission Rates and Changes of Leukemia Stem Cells
Brief Title: Pegylated Liposomal Doxorubicin Versus Daunorubicin to Treat Acute Lymphoblastic Leukemia:
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changzhou Jinyuan Pharmaceutical Manufacturing Co., Ltd. (Other)
Collaborators: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChangzhouJP
Record Dates: First submitted 2014-02-20; First posted 2014-02-25 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-02

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PLD-contained VDCLD regimen (Experimental): PLD 36 mg/m2 ivdrip over 60 minutes( d1、15),VCR 1.4mg/m iv(d1，8，15，22), CTX 800 mg/m2 ivdrip( d1), L-asp 6000u/m2 ivdrip(d19～28),Dex10mg ivdrip (d1～28).
  Interventions: Drug: VDCLD regimen
- DNR-contained VDCLD regimen (Active Comparator): DNR 45 mg/m2 ivdrip over 60 minutes(d1～3),VCR 1.4mg/m2 iv(d1，d8，d15，d22), CTX 800 mg/m2 ivdrip(d1), L-asp 6000u/m2 ivdrip(d19～28),Dex10mg ivdrip(d1～28).
  Interventions: Drug: VDCLD regimen

INTERVENTIONS:
Drug: VDCLD regimen

SUMMARY:
To determine, compared with Daunorubicin(DNR), whether Pegylated liposomal doxorubicin (PLD) inducing higher complete remission (CR) rate, in untreated primary ALL adult patients with VDCLD regimen induction therapy. Second, to determine, compared with the DNR, whether chemotherapy containing PLD with a higher response rates and greater safety in adult ALL

DETAILED DESCRIPTION:
This is a prospective, multicenter, open, non-intervention clinical study, with estimated enrollment of 200 newly diagnosed adult ALL patients. After the first course of treatment administered with PLD-contained or DNR-contained VDCLD regimen, CR rate and changes of leukemia stem cells in bone marrow, was evaluated; the safety of these chemotherapy was also evaluated.

Study Patients:

Patients included in this study should be untreated with ALL previously, being in line with the inclusion criteria and exclusion criteria.

Dosage and Administration:

PLD-contained VDCLD regimen：PLD 36 mg/m2 ivdrip over 60 minutes( d1、15),VCR 1.4mg/m iv(d1，8，15，22), CTX 800 mg/m2 ivdrip( d1), L-asp 6000u/m2 ivdrip(d19～28),Dex10mg ivdrip (d1～28).

DNR-contained VDCLD regimen：DNR 45 mg/m2 ivdrip over 60 minutes(d1～3),VCR 1.4mg/m2 iv(d1，d8，d15，d22), CTX 800 mg/m2 ivdrip(d1), L-asp 6000u/m2 ivdrip(d19～28),Dex10mg ivdrip(d1～28).

Endpoints:

Primary endpoint: The primary endpoint of the study was complete remission (CR) rates after the first course of regimen. The proportion of patients achieved CR was evaluated, after the first course of induction chemotherapy administered with PLD-contained or DNR-contained VDCLD regimen Secondary endpoint: The change of leukemia stem cells in bone marrow, was evaluated before and after administered with PLD-contained or DNR-contained VDCLD regimen.

Safety Assessment:

In order to adjust the treatment strategy and ensure patients' safety effectively, routine blood test, transaminases, and creatinine was monitored on time during the period, while lung CT and ECG was performed based on clinical need. Possible adverse reactions and tolerability during treatment, such as gastrointestinal reactions, cardiac function, as well as discontinuation ratio due to side effects or tolerability of PLD, was recorded.

Statistical Analysis:

All the calculations were performed with the SPSS statistical software. The continuous variables were performed with T test; categorical variables were performed withχ2 test. After acceptance of various observation records sheets, data were unified processed.

ELIGIBILITY:
Inclusion Criteria:

Eligible men or women were age over 14，but less than 60 years;

Eastern Cooperative Oncology Group performance status of 0 to2;

Diagnosed with ALL (WHO classification, the primitive cells ≥ 20%);

Previous untreated ALL patients had not received chemotherapy before (excluding dexamethasone, prednisone, and hydroxyurea). History of receiving blood transfusion, hematopoietic growth factors, vitamin, and palliative measures such as leukocyte removal, dexamethasone, prednisone, hydroxyurea (0.5-3g daily, more than three days) is allowed;

The levels of LSCs in bone marrow were measured with flow cytometry before treatment;

Subjects must be able to provide written informed consent.

Exclusion Criteria:

Mixed type of AL patients;

Clinically significant active infections;

Nursing (breastfeeding) or intending to be nursing during the study；

Pregnancy, or intending to become pregnant during the study;

Patients with cardiac dysfunction currently (especially congestive heart failure) or history of congestive heart failure;

Patients with severe liver failure (ALT ≥ 5 times the upper limit of normal (ULN), total bilirubin ≥ 3mg/dL)

Patients with renal insufficiency, creatinine clearance <30ml/min, creatinine clearance rate is calculated as follows: Men: Ccr (ml / min) = (140 - age) × weight (kg) / [0.8136 × serum creatinine (μmol / L )] female: Ccr (ml / min) = (140 - age) × weight (kg) × 0.85 / [0.8136 × serum creatinine (μmol / L)];

Patients did not or will not participate in other trials of drugs 30 days before or 90 days after the beginning of this study,

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) rates after the first course of regimen | 3 years after the last enrollment
  The primary endpoint of the study was complete remission (CR) rates after the first course of regimen. The proportion of patients achieved CR was evaluated, after the first course of induction chemotherapy administered with PLD-contained or DNR-contained VDCLD regimen

SECONDARY OUTCOMES:
The change of leukemia stem cells in bone marrow | 3 years after the last enrollment
  The change of leukemia stem cells in bone marrow, was evaluated before and after administered with PLD-contained or DNR-contained VDCLD regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Zhigang Yang, Principal Investigator — Affiliated Hospital of Guangdong Medical University
Locations (1):
- Department of Hematology, Affiliated Hospital of Guangdong Medical College, Zhanjiang, Guangdong, China